CLINICAL TRIAL: NCT00429273
Title: An Eight-Week, Randomized, Double-Blind Comparison of Guanfacine, Focalin XR, and the Combination, With a Twelve Month Open-Label Extension for the Treatment of ADHD in Pediatric Subjects Aged 7 to 14 Years
Brief Title: Single Versus Combination Medication Treatment for Children With Attention Deficit Hyperactivity Disorder
Acronym: Project1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, James McCracken, Chair, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P50MH077248-01 (NIH); P50MH077248-01 (NIH); 10-000453 (Other: Office for Protection of Human Subjects)
Record Dates: First submitted 2007-01-29; First posted 2007-01-31 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: ADHD; Guanfacine; Methylphenidate; Focalin XR; Pediatric; Cognitive function; Combination therapy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Guanfacine; Methylphenidate; Dexmethylphenidate Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1: Guan-Guan+Placebo (Active Comparator): weeks 1-4: Guanfacine weeks 5-8: Guanfacine + Placebo
  Interventions: Drug: Guanfacine
- Group 2: Placebo-Placebo+DMPH (Active Comparator): weeks 1-4: Placebo weeks 5-8: Placebo+DMPH
  Interventions: Drug: Methylphenidate (MPH)
- Group 3: Guan-Guan+DMPH (Comb) (Experimental): weeks 1-4: Guanfacine weeks 5-8: Guanfacine+DMPH
  Interventions: Drug: Guanfacine; Drug: Methylphenidate (MPH)

INTERVENTIONS:
Drug: Guanfacine — Week 1: 0.5 mg twice daily; Week 2: 1 mg twice daily; Week 3: 1.5 mg twice daily; Weeks 4 through 8: best dose as determined by efficacy measures
  Other Names: Tenex
  Arms: Group 1: Guan-Guan+Placebo; Group 3: Guan-Guan+DMPH (Comb)
Drug: Methylphenidate (MPH) — Participants less than 25 kg will receive 10 mg once daily for Week 5, 20 mg once daily for Week 6, and 30 mg once daily for Week 7. Subjects greater than 25 kg will receive 20 mg once daily for Week 5, 30 mg once daily for Week 6, 40 mg once daily for Week 7, and best doses as determined by efficacy measures for Week 8.
  Other Names: Focalin XR
  Arms: Group 2: Placebo-Placebo+DMPH; Group 3: Guan-Guan+DMPH (Comb)

SUMMARY:
This study will evaluate the effectiveness of a single drug versus a combination of drugs in treating attention deficit hyperactivity disorder in children.

DETAILED DESCRIPTION:
Attention deficit hyperactivity disorder (ADHD) is one of the most common childhood mental disorders. Children with ADHD have impaired functioning in multiple settings, including home and school. They also have difficulty relating with peers. If left untreated, the disorder may cause adverse effects that can last into adolescence and adulthood. Stimulant medications, such as methylphenidate, are effective in reducing ADHD symptoms on a short-term basis. However, few long-term benefits in academic or general functioning from current ADHD therapies have been demonstrated. Focalin XR is a stimulant medication that is FDA-approved for treating ADHD. Guanfacine is another medication that is currently approved for the treatment of hypertension, but has long been used for treating ADHD. This study will determine the effectiveness of a combination of Focalin XR and guanfacine in enhancing cognitive functioning and improving the long-term benefit of ADHD treatment.

Participants in this study will be randomly assigned to one of three treatment regimens: Methylphenidate (Focalin XR) and placebo; guanfacine and placebo; or Focalin XR and guanfacine. The study will be conducted in two phases: an 8-week double-blind treatment phase and a 12-month open-label treatment phase. In Phase I, one third of participants will receive placebo for the initial 4 weeks, followed by Focalin XR alone for the remaining 4 weeks. All other participants will receive their assigned medications for the full 8 weeks. All participants will attend two study visits prior to beginning treatment and one study visit per week throughout Phase I. At the end of Phase I, treatment assignments will be unblinded. Participants who experienced adequate improvement with their assigned treatment will then continue in Phase II on the same medication(s) for an additional 12 months. Participants will attend study visits once per month until the end of the study. Study visits will include self-report measures, clinical assessments, and cognitive testing. Participants will also undergo four electroencephalography (EEG) tests and two fMRI scans over the course of the study. All Phase II participants will receive a follow-up telephone call 1 month after the final study visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DSM-IV ADHD by K-SADS-PL and confirmed by clinical interview
* Clinical Global Impression-Severity score of at least 4 for ADHD
* Resided with primary caretaker for at least 6 months prior to study entry

Exclusion Criteria:

* History of autism, pervasive developmental disorder, chronic tic disorder, psychosis, or bipolar disorder
* Current major depression or panic disorder
* Systolic or diastolic blood pressure at screening greater than the 95th percentile or less than the 5th percentile for age and body mass index (BMI)
* Any medical condition that might make stimulant or alpha agonist therapy medically inadvisable
* Need for chronic use of other medications with central nervous system effects
* Pregnant, breastfeeding, or beyond menarche and has a positive urine pregnancy test
* History of structural heart defects, syncope, or fainting while exercising
* Clinically significant cardiac abnormality as determined by echocardiogram (ECG) at study entry
* Mental retardation as determined by clinical functional assessment and an IQ estimate of less than 70 based on Wechsler Adult Intelligence Scale (WAIS) subtests

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 212 (Actual)
Dates: Start 2007-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James T. McCracken, MD, Principal Investigator — University of California, Los Angeles; James J. McGough, MD, Study Director — University of California, Los Angeles
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Storebo OJ, Storm MRO, Pereira Ribeiro J, Skoog M, Groth C, Callesen HE, Schaug JP, Darling P, Huus CL, Zwi M, Kirubakaran R, Simonsen E, Gluud C. Methylphenidate for children and adolescents with attention deficit hyperactivity disorder (ADHD). Cochrane Database Syst Rev. 2025 Dec 4;12(12):CD009885. doi: 10.1002/14651858.CD009885.pub4. PMID 41342306
- [Derived] Storebo OJ, Storm MRO, Pereira Ribeiro J, Skoog M, Groth C, Callesen HE, Schaug JP, Darling Rasmussen P, Huus CL, Zwi M, Kirubakaran R, Simonsen E, Gluud C. Methylphenidate for children and adolescents with attention deficit hyperactivity disorder (ADHD). Cochrane Database Syst Rev. 2023 Mar 27;3(3):CD009885. doi: 10.1002/14651858.CD009885.pub3. PMID 36971690
- [Derived] Michelini G, Lenartowicz A, Vera JD, Bilder RM, McGough JJ, McCracken JT, Loo SK. Electrophysiological and Clinical Predictors of Methylphenidate, Guanfacine, and Combined Treatment Outcomes in Children With Attention-Deficit/Hyperactivity Disorder. J Am Acad Child Adolesc Psychiatry. 2023 Apr;62(4):415-426. doi: 10.1016/j.jaac.2022.08.001. Epub 2022 Aug 10. PMID 35963559
- [Derived] Michelini G, Lenartowicz A, Diaz-Fong JP, Bilder RM, McGough JJ, McCracken JT, Loo SK. Methylphenidate, Guanfacine, and Combined Treatment Effects on Electroencephalography Correlates of Spatial Working Memory in Attention-Deficit/Hyperactivity Disorder. J Am Acad Child Adolesc Psychiatry. 2023 Jan;62(1):37-47. doi: 10.1016/j.jaac.2022.06.017. Epub 2022 Aug 10. PMID 35963558
- [Derived] Sayer GR, McGough JJ, Levitt J, Cowen J, Sturm A, Castelo E, McCracken JT. Acute and Long-Term Cardiovascular Effects of Stimulant, Guanfacine, and Combination Therapy for Attention-Deficit/Hyperactivity Disorder. J Child Adolesc Psychopharmacol. 2016 Dec;26(10):882-888. doi: 10.1089/cap.2015.0264. Epub 2016 Aug 2. PMID 27483130
- [Derived] Loo SK, Bilder RM, Cho AL, Sturm A, Cowen J, Walshaw P, Levitt J, Del'Homme M, Piacentini J, McGough JJ, McCracken JT. Effects of d-Methylphenidate, Guanfacine, and Their Combination on Electroencephalogram Resting State Spectral Power in Attention-Deficit/Hyperactivity Disorder. J Am Acad Child Adolesc Psychiatry. 2016 Aug;55(8):674-682.e1. doi: 10.1016/j.jaac.2016.04.020. Epub 2016 May 21. PMID 27453081
- [Derived] Bilder RM, Loo SK, McGough JJ, Whelan F, Hellemann G, Sugar C, Del'Homme M, Sturm A, Cowen J, Hanada G, McCracken JT. Cognitive Effects of Stimulant, Guanfacine, and Combined Treatment in Child and Adolescent Attention-Deficit/Hyperactivity Disorder. J Am Acad Child Adolesc Psychiatry. 2016 Aug;55(8):667-73. doi: 10.1016/j.jaac.2016.05.016. Epub 2016 Jun 7. PMID 27453080
- [Derived] McCracken JT, McGough JJ, Loo SK, Levitt J, Del'Homme M, Cowen J, Sturm A, Whelan F, Hellemann G, Sugar C, Bilder RM. Combined Stimulant and Guanfacine Administration in Attention-Deficit/Hyperactivity Disorder: A Controlled, Comparative Study. J Am Acad Child Adolesc Psychiatry. 2016 Aug;55(8):657-666.e1. doi: 10.1016/j.jaac.2016.05.015. Epub 2016 Jun 3. PMID 27453079

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 212 randomized (deemed eligible and enrolled). 71 randomized to Group 1: 3 dropped prior to receiving drug; thus 68 started drug.
  70 randomized to Group 2: 1 dropped before receiving drug; thus 69 started drug.
  71 randomized to Group 3:1 dropped before receiving drug; thus 70 started drug.
Groups:
- Group 1: Guan-Guan+Placebo: weeks 1-4: Guanfacine weeks 5-8: Guanfacine+Placebo
- Group 3: Guan-Guan+DMPH: weeks 1-4: Guanfacine weeks 5-8: Guanfacine+DMPH (comb)
Period: Overall Study
Arm/Group | Group 1: Guan-Guan+Placebo | Group 2: Placebo-Placebo+DMPH | Group 3: Guan-Guan+DMPH
Started | 68 | 69 | 70
Completed | 60 | 61 | 61
Not Completed | 8 | 8 | 9
Not completed — Lost to Follow-up | 1 | 2 | 2
Not completed — Physician Decision | 6 | 5 | 5
Not completed — Adverse Event | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Guan-Guan+Placebo: weeks 1-4: Guanfacine weeks 5-8: Guanfacine +Placebo
- Group 3: Guan-Guan+DMPH (Comb): weeks 1-4: Guanfacine weeks 5-8: Guanfacine+DMPH (comb)
- Total: Total of all reporting groups
Arm/Group | Group 1: Guan-Guan+Placebo | Group 2: Placebo-Placebo+DMPH | Group 3: Guan-Guan+DMPH (Comb) | Total
Number analyzed (Participants) | 68 | 69 | 70 | 207
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.1 (2.1) | 10.1 (2.0) | 9.9 (2.2) | 10.0 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 19 | 65
  Male | 45 | 46 | 51 | 142
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: of the 212 participants randomized, 207 received at least one dose of study drug and form the safety and intent-to-treat samples.
  Participants
    White | 51 | 51 | 41 | 143
    African American | 7 | 10 | 19 | 36
    Asian, Pacific Islander | 7 | 4 | 5 | 16
    Other | 3 | 4 | 5 | 12
    Hispanic | 16 | 10 | 18 | 44

OUTCOME MEASURES:

1. Primary Outcome: ADHD IV Rating Scale (Attention Deficit Hyperactivity Disorder Rating Scale)
Description: The primary clinical efficacy variable for treatment was the ADHD-RS-IV (Attention-Deficit/Hyperactivity Disorder Rating Scale) Total Score and two sub-scales (Inattentive and Hyperactive-Impulsive ).
  The rating scale has 18 questions with answer options: None (0), Mild (1), Moderate (2) and Severe (3). Min 0; max 3.
  Scores are obtained by summing each item; The higher the score, the worse the outcome.
  Total score range: 0-54 Total Inattentive score range: 0-27 Total Hyperactive/Impulsive score range: 0-27
Time Frame: Measured at baseline Week 4 and Week 8
Population: Every contrast includes estimates of maturation/time trend and the within subject covariance structure based on all participants using full information maximum likelihood estimation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Estimated Difference Between Guan and Placebo: Contrasts based on all observations of patients treated with guam and all patients on placebo controlling for time effects. For placebo this included patients in the guan-guan arm at baseline, the guan-combo arm at baseline, and the placebo-DMPH arm at baseline and 4 weeks, while the estimates for guan are based on the guan-guan arm both at 4 weeks and 8 weeks, and the guan-combo arm at 4 weeks only. Participant specific effects and time effects are controlled for based on estimates from all participants and all time points.
- Estimated Difference Between DMPH and Placebo: Contrasts based on all observations of patients treated with dmph and all patients on placebo controlling for time effects. For placebo this included patients in the guan-guan arm at baseline, the guan-combo arm at baseline, and the placebo-DMPH arm at baseline and 4 weeks, while the estimates for DMPH are based on the placebo-guan arm at 8 weeks. Participant specific effects and time effects are controlled for based on estimates from all participants and all time points.
- Estimated Difference Between Placebo and Combo: Contrasts based on all observations of patients treated with combo and all patients on placebo controlling for time effects. For placebo this included patients in the guan-guan arm at baseline, the guan-combo arm at baseline, and the placebo-DMPH arm at baseline and 4 weeks, while the estimates for DMPH are based on the guan-combo arm at 8 weeks. Participant specific effects and time effects are controlled for based on estimates from all participants and all time points.
Arm/Group | Estimated Difference Between Guan and Placebo | Estimated Difference Between DMPH and Placebo | Estimated Difference Between Placebo and Combo
Number analyzed (Participants) | 207 | 207 | 207
units on a scale
  Total ADHD-RS Score | -7.77 (1.70) | -7.99 (1.22) | -10.66 (1.99)
  Inattentive Subscale | -4.14 (0.99) | -4.10 (0.71) | -5.89 (1.15)
  Hyperactive Impulsive Subscale | -3.73 (0.92) | -4.0 (0.69) | -5.10 (1.12)
Statistical Analysis 1: Comparison: Estimated Difference Between Guan and Placebo vs Estimated Difference Between DMPH and Placebo vs Estimated Difference Between Placebo and Combo; Analyses are based on a generalized linear mixed model (GLMM) modelling the effects of the medication when calibrated to optimal dosage and controlling for time effects and within-subject effects. The design is a combined within-between subject design, where each participant is exposed to, and provides information about multiple tx modalities; Test type: Other — Test for differences in treatment outcomes between three different tx; p < .01, Mixed Models Analysis; F-Value for variance component = 18.90

ADVERSE EVENTS:
Groups:
- Group 1: Guan-Guan+Placebo: week 1-4: Guanfacine weeks 5-8: Guanfacine+Placebo
- Group 2: Placebo-Placebo+DMPH: week 1-4: Placebo week 5-8: Placebo+DMPH
- Group 3: Guan-Guan+DMPH: week 1-4: Guanfacine week 5-8: Guanfacine+DMPH (comb)
Arm/Group | Group 1: Guan-Guan+Placebo | Group 2: Placebo-Placebo+DMPH | Group 3: Guan-Guan+DMPH
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/69 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/69 | 0/70
Other Adverse Events (participants affected / at risk) | 66/68 | 66/69 | 69/70
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Guan-Guan+Placebo (N=68) | Group 2: Placebo-Placebo+DMPH (N=69) | Group 3: Guan-Guan+DMPH (N=70)
Abdominal Pain Upper (Gastrointestinal disorders) | 11 (11) | 10 (10) | 10 (10)
Abdominal Pain (Gastrointestinal disorders) | 19 (19) | 18 (18) | 16 (16)
Headache (Psychiatric disorders) | 34 (34) | 23 (23) | 23 (23)
Irritability (Psychiatric disorders) | 15 (15) | 12 (12) | 18 (18)
Sedation (Psychiatric disorders) | 12 (12) | 4 (4) | 16 (16)
Somnolence (Psychiatric disorders) | 16 (16) | 3 (3) | 15 (15)
Affect Lability (Psychiatric disorders) | 7 (7) | 14 (14) | 8 (8)
Insomnia (General disorders) | 18 (18) | 20 (20) | 24 (24)
Decreased Appetite (Metabolism and nutrition disorders) | 15 (15) | 31 (31) | 25 (25)
Lethargy (General disorders) | 23 (23) | 9 (9) | 16 (16)
Fatigue (General disorders) | 22 (22) | 5 (5) | 12 (12)
Dizziness (Vascular disorders) | 8 (8) | 6 (6) | 7 (7)

LIMITATIONS AND CAVEATS:
Larger group sizes would enable more conclusive tests of treatment differences; Study design began with guanfacine first and addition of a stimulant second, making difficult to compare to those study designs adding guanfacine to ongoing stimulants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No